CLINICAL TRIAL: NCT07389824
Title: Efficacy of Acupuncture Combined With Mesalazine in Inducing and Maintaining Clinical Remission in Mild-to-Moderate Active Ulcerative Colitis: A Single-Center, Randomized Controlled Clinical Trial.
Brief Title: Efficacy of Acupuncture-Mesalazine Combination Therapy in Ulcerative Colitis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qin Yu (Other)
Responsible Party: Sponsor-Investigator, Qin Yu, Associate Professor, Chief Physician, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UC-ACU(2025TJ01)
Record Dates: First submitted 2026-01-02; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: Acupuncture; Mesalazine; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Acupuncture Therapy; Mesalamine

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups in a 1:1 ratio.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum acupuncture (Experimental): Participants receive intradermal thumbtack needle embedding at four fixed acupoints (bilateral BL25 and ST36) and one optional pair selected from ST25 (for damp-heat), BL20 (for spleen deficiency/dampness), BL23 (for spleen-kidney yang deficiency), or SP6 (for liver depression/spleen deficiency) based on TCM pattern diagnosis. Needles are embedded for up to 72 hours; patients press them 3-5 times daily to elicit deqi sensation. Needles are replaced weekly for 12 weeks. All participants concurrently receive standard mesalazine therapy.
  Interventions: Device: Acupuncture; Drug: Mesalazine
- sham acupuncture (Sham Comparator): Participants receive sham acupuncture using needle-free adhesive placebo patches (identical in appearance to verum needles) applied at two fixed pairs of non-acupoints (4 points total), away from true meridians or acupoints. Patients are instructed to apply gentle pressure to the patch sites 3-5 times daily , without eliciting deqi sensation. Patches are replaced weekly for 12 consecutive weeks. All participants concurrently receive standard mesalazine therapy.
  Interventions: Device: Sham acupuncture; Drug: Mesalazine

INTERVENTIONS:
Device: Acupuncture — Intradermal thumbtack needle embedding at specified acupoints. Needles are embedded for up to 72 hours, replaced weekly for 12 weeks. Patients press needles 3-5 times daily to elicit deqi sensation.
  Other Names: Acupuncture with intradermal thumbtack needle
  Arms: Verum acupuncture
Device: Sham acupuncture — Application of needle-free adhesive placebo patches at non-acupoint sites. Patches are replaced weekly for 12 weeks. Patients apply gentle pressure 3-5 times daily without deqi sensation.
  Other Names: Sham acupuncture with sham intradermal thumbtack needle
  Arms: sham acupuncture
Drug: Mesalazine — Standard background therapy: Mesalazine at a stable dose (e.g., 2-4g/day) maintained throughout the 12-week study period. This provides the background treatment for both groups, allowing evaluation of the additive effect of acupuncture.
  Other Names: 5-ASA; 5-aminosalicylic acid

SUMMARY:
This study aims to evaluate the efficacy and safety of acupuncture combined with mesalazine (an integrated acupuncture-medication regimen) for ulcerative colitis.

DETAILED DESCRIPTION:
1. A randomized controlled trial.
2. Acupuncture treatment(intradermal thumbtack needle embedding), placebo control.
3. To explore the efficacy and safety of acupuncture(intradermal thumbtack needles embedding) as an adjuvant therapy for active ulcerative colitis.
4. To explore the potential relevant mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. documented diagnosis of UC；
2. age 18-65 years, regardless of gender;
3. mildly to moderately active UC, defined as a baseline total Mayo score between 3 and 10；
4. willing to receive the complete protocol of intradermal thumbtack needle embedding therapy (12 sessions across three treatment courses)；
5. Willing to undergo two colonoscopies (pre-treatment and post-treatment)；
6. complete all baseline assessments;
7. capable of understanding and voluntarily sign the informed consent form.

Exclusion Criteria:

1. diagnosed with or suspected to have other type of inflammatory bowel disease, such as Crohn's disease;
2. patients in clinical remission or with severe disease activity ( baseline total Mayo score < 3, or > 10 );
3. having severe gastrointestinal complications or a recent surgical history, including but not limited to: short bowel syndrome, toxic megacolon, intestinal perforation, complete intestinal obstruction, active massive gastrointestinal hemorrhage, or having undergone major abdominal or intestinal surgery within the past 6 months.
4. patients unwilling to undergo colonoscopy;
5. significant or unstable comorbidities (e.g., cardiovascular, respiratory, hepatic, or renal diseases);
6. patients with malignant tumors (including but not limited to colorectal cancer);
7. patients with a history of intradermal thumbtack needle embedding;
8. pregnant or lactating women;
9. patients with mental illness;
10. patients with either coagulation disorders or skin conditions (such as diseases, infections, ulcers, scars, or tumors at the acupuncture sites) that would preclude acupuncture；
11. strong needle phobia or unwillingness to receive acupuncture treatment;
12. any other condition (e.g., geographical remoteness, history of poor adherence) that, in the opinion of the investigator, would make the patient unsuitable for the study or likely to be non-compliant with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate | Week 13-16 after randomization
  Proportion of patients who achieve a Mayo Stool Frequency Subscore (SFS) of 0 or 1 and not increased from induction baseline, a Mayo Rectal Bleeding Subscore (RBS) of 0, and a Mayo Endoscopic Score(MES) of 0 or 1 with no friability present on endoscopy.

SECONDARY OUTCOMES:
Clinical response rate | Week 13-16 after randomization
  Proportion of patients with a decrease from induction baseline in the mMayo score by at least 30% and at least 2 points, with either a 1-point or more decrease from induction baseline in the Mayo Rectal Bleeding Subscore (RBS) or a Mayo RBS of 0 or 1
Endoscopic improvement rate | Week 13-16 after randomization
  Proportion of patients with a Mayo Endoscopic Subscore (MES) of 0 or 1 (no friability) or an Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score of 0 or 1.
Endoscopic remission (normalization) rate | Week 13-16 after randomization
  Proportion of patients with a Mayo Endoscopic Subscore (MES) of 0.
Symptomatic remission rate | Week 12 and 24 after randomization
  Proportion of patients with a Mayo Stool Frequency Subscore (SFS) of 0 or 1 and not increased from induction baseline, and a Mayo Rectal Bleeding Subscore (RBS) of 0
Symptomatic response rate | Week 12 and 24 after randomization
  Proportion of patients with a decrease from baseline in the symptomatic Mayo score (SFS+RBS) by ≥30% and ≥1 point, plus either a ≥1-point decrease in RBS or an RBS of 0 or 1.
Number of remission-relapse episodes | Week 24 after randomization
  Incidence of clinical recurrences(defined per STRIDE-II consensus) within 24 weeks post-randomization.
Time to first relapse | Week 24 after randomization
  Time to first relapse within 24 weeks post-randomization
Use of rescue medication | Week 24 after randomization
  Proportion of patients requiring glucocorticoids, immunosuppressants, biologics, or other rescue medications due to disease progression.
Change in Nancy Histological Index score | Week 13-16 after randomization
  Change from baseline in the Nancy Histological Index score, a validated scale for assessing histological disease activity in ulcerative colitis, with scores ranging from 0 (no activity) to 3 (severe activity). A higher score indicates more severe histological inflammation.
Change in fecal calprotectin level | Baseline, Week 12, Week 24
  Change from baseline in fecal calprotectin concentration
Change in C-reactive protein level | Baseline, Week 12, Week 24
  Change from baseline in serum C-reactive protein (CRP) concentration.
Change in erythrocyte sedimentation rate | Baseline, Week 12, Week 24
  Change from baseline in erythrocyte sedimentation rate (ESR).
Change in hemoglobin level | Baseline, Week 12, Week 24
  Change from baseline in hemoglobin (Hb) concentration.
Change in Inflammatory Bowel Disease Questionnaire (IBDQ) score | Baseline, Week 12, Week 24
  Change from baseline in the total score of the Inflammatory Bowel Disease Questionnaire (IBDQ). The IBDQ is a 32-item questionnaire measuring quality of life in IBD patients, with total scores ranging from 32 to 224. A higher score indicates a better quality of life.
Change in Pittsburgh Sleep Quality Index (PSQI) score | Baseline, Week 12, Week 24
  Change from baseline in the global score of the Pittsburgh Sleep Quality Index (PSQI). The PSQI assesses sleep quality over a 1-month interval, with global scores ranging from 0 to 21. A higher score indicates worse sleep quality.
Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) score | Baseline, Week 12, Week 24
  Change from baseline in the score of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) subscale. The FACIT-Fatigue is a 13-item subscale measuring fatigue, with scores ranging from 0 to 52. A higher score indicates less fatigue (better outcome).
Change in Beck Depression Inventory-II (BDI-II) score | Baseline, Week 12, Week 24
  Change from baseline in the total score of the Beck Depression Inventory-II (BDI-II). The BDI-II is a 21-item self-report inventory measuring the severity of depression, with total scores ranging from 0 to 63. A higher score indicates more severe depressive symptoms.
Change in Beck Anxiety Inventory (BAI) score | Baseline, Week 12, Week 24
  Change from baseline in the total score of the Beck Anxiety Inventory (BAI). The BAI is a 21-item self-report inventory measuring the severity of anxiety, with total scores ranging from 0 to 63. A higher score indicates more severe anxiety symptoms.
De Qi sensation on the Massachusetts General Hospital Acupuncture Sensation Scale (MASS) | Week 12 after randomization
  Score on the Massachusetts General Hospital Acupuncture Sensation Scale (MASS), a validated instrument assessing 12 sensations associated with De Qi (e.g., soreness, numbness, distension). The total score is a weighted sum, with a higher score indicating a more pronounced De Qi experience.
Change in Acupuncture Treatment Expectancy score | Baseline, Week 12 after randomization
  Change from baseline in the score of the Acupuncture Expectancy Scale (AES), a questionnaire assessing patients' belief in the potential benefit of acupuncture treatment. A higher score indicates greater treatment expectancy.
Incidence of acupuncture-related adverse events | Throughout the 12-week treatment period
  Number and percentage of participants experiencing any acupuncture-related adverse event (e.g., local hematoma, intense pain [VAS ≥8], infection) or other discomfort (e.g., nausea, dizziness) following each acupuncture session, assessed over the entire treatment period.
Change in abdominal symptoms severity score | Week 24 after randomization
  Change from baseline in the severity of abdominal symptoms (including defecation urgency and abdominal pain) as assessed by a Numerical Rating Scale (NRS). The NRS is a self-report scale ranging from 0 ("no symptom") to 10 ("worst imaginable symptom"). A higher score indicates more severe symptoms.
Change in Patient-Doctor Relationship Questionnaire (PDRQ-9) score | Baseline, Week 12, Week 24
  Change from baseline in the total score of the Patient-Doctor Relationship Questionnaire (PDRQ-9). The PDRQ-9 is a 9-item questionnaire assessing the quality of the patient-doctor relationship, with total scores ranging from 9 to 45. A higher score indicates a better perceived relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Qin, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
IPD after de-identification can be shared on individual request to the principal investigator at yuqin@tjh.tjmu.edu.cn
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available after the publication of the primary outcomes
Access Criteria: Data requests from qualified researchers for the purpose of replicating analyses or conducting secondary analyses will be considered. Requestors must submit a research proposal outlining the scientific purpose and analysis plan to the principal investigator via the contact email. Approval will be granted based on scientific merit, feasibility, and adherence to data use agreements.